CLINICAL TRIAL: NCT00353795
Title: Coronary Atherosclerosis Evaluation by Arterial Wall MRI
Brief Title: Coronary Atherosclerosis Evaluation by Arterial Wall Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Northwestern University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-05-23-01; 5R01HL078909 (NIH)
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Arteriosclerosis; Arteriosclerosis, Coronary; Atherosclerosis, Coronary; Coronary Artery Disease; Coronary Atherosclerosis
Keywords: MESA; MRI; Cardiovascular; Cardiac; Coronary; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

INTERVENTIONS:
Procedure: MR Imaging of the Coronary Arteries

SUMMARY:
The overall goal of this study is to use MRI to:

* Examine the relationship between known risk factors for cardiovascular disease and coronary artery wall thickness;
* Examine the relationship between coronary artery wall thickness and other markers of subclinical coronary atherosclerosis, such as carotid wall thickness and coronary calcium scores; and,
* Examine the feasibility of measuring the progression of coronary artery wall thickness over time in a subset of participants.

DETAILED DESCRIPTION:
Each enrolled participant will undergo MR Imaging of the coronary arteries in conjunction with their routine MESA follow-up visit. The MRI will last approximately 45-60 minutes

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in the MESA Study at the Hopkins MESA Field Center or the Northwestern University MESA Field Center
* Male or Female adult equal to or older than 45 years of age
* Willing/able to provide informed consent

Exclusion Criteria:

* Any known contraindications to MRI (i.e. severe claustrophobia, pacemaker, etc.)
* Metal in the eyes

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Bluemke, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Northwestern University MESA Field Center, Chicago, Illinois
  - Johns Hopkins MESA Field Center, Baltimore, Maryland

REFERENCES:
- See also: Multi-Ethnic Study of Atherosclerosis webpage — http://www.mesa-nhlbi.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Participants in the MESA trial (http://www.mesa-nhlbi.org/) randomly selected by the University of Washington Coordinating center who agreed to participate. Enrollment from October 2005 to February 2008
Period: Overall Study
Arm/Group | Participants
Started | 179
Completed | 179
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 179
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 89
Region of Enrollment [Number; unit: participants]
  United States | 179

OUTCOME MEASURES:

1. Primary Outcome: Mean Coronary Wall Thickness
Description: Average thickness of the wall of the left anterior descending, right and left main coronary artery measured by magnetic resonance imaging (MRI).
Time Frame: n/a (cross sectional analysis)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Participants
Number analyzed (Participants) | 179
mm | 2.0 (0.3)

ADVERSE EVENTS:
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 0/179
Other Adverse Events (participants affected / at risk) | 0/179

LIMITATIONS AND CAVEATS:
Cross sectional study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes